CLINICAL TRIAL: NCT07194447
Title: The Effect of Locally Applied Gel-Based Simvastatin on Dental Implant Stability and Marginal Bone Level : A Randomized Controlled Double-Blind Clinical Trial
Brief Title: Effect of Locally Applied Simvastatin Gel on Dental Implant Stability and Marginal Bone Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maha Zuhair (Other)
Responsible Party: Sponsor-Investigator, Maha Zuhair, Maha Zuhair Ahmed Al-Chalabi, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UBaghdad-ImplantSIMV-2025
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Dental Implants , Osseointegration , Marginal Bone Loss , Implant Stability
Keywords: Simvastatin, Local Drug Delivery, Dental Implant Stability , Marginal Bone Level , ,

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1 ratio to either the test group (simvastatin gel) or the control group (methylcellulose gel).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind design was implemented to ensure that participants, care providers, investigators, and outcome assessors were unaware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simvastatin Gel Group (Active Comparator): Participants received dental implants with a single local application of 1.2% simvastatin in 4% methylcellulose gel applied around the implant site immediately after implant placement and prior to flap closure.
  Interventions: Drug: Simvastatin Gel
- Control Gel Group (Placebo Comparator): articipants received dental implants with a single local application of 4% methylcellulose gel without simvastatin, applied around the implant site immediately after implant placement and prior to flap closure.
  Interventions: Drug: Methylcellulose Gel

INTERVENTIONS:
Drug: Simvastatin Gel — A single local application of 1.2% simvastatin incorporated into 4% methylcellulose gel, placed around the implant site immediately after implant placement and before flap closure.
  Arms: Simvastatin Gel Group
Drug: Methylcellulose Gel — A single local application of 4% methylcellulose gel without simvastatin, placed around the implant site immediately after implant placement and before flap closure.
  Arms: Control Gel Group

SUMMARY:
stability and marginal bone level. Forty-two patients received dental implants and were randomly assigned to two groups. In the test group, 1.2% simvastatin in 4% methylcellulose gel was applied around the implant, while in the control group, methylcellulose gel alone was used. Implant stability was measured using resonance frequency analysis at baseline, 8 weeks, and 16 weeks. Marginal bone level was assessed by cone-beam computed tomography (CBCT) at baseline and 16 weeks. The aim of the study was to investigate whether local application of simvastatin enhances osseointegration and reduces marginal bone loss compared to the control treatment.

DETAILED DESCRIPTION:
ental implant stability is a key factor for the long-term success of implant therapy. Stability depends initially on primary mechanical fixation and later on secondary biological osseointegration. Various pharmacological agents have been suggested to promote bone formation around implants, including statins. Statins, primarily used as lipid-lowering agents, also demonstrate pleiotropic effects, such as stimulating bone morphogenetic protein-2 (BMP-2) expression and enhancing osteoblastic differentiation.

This randomized, double-blind, controlled clinical trial was designed to evaluate the effect of locally applied simvastatin gel on implant stability and marginal bone level. A total of 42 patients requiring single dental implants were enrolled. Participants were randomly allocated into two groups:

Simvastatin group (test): Implants placed with local application of 1.2% simvastatin in 4% methylcellulose gel.

Control group: Implants placed with local application of 4% methylcellulose gel only.

Implant stability quotient (ISQ) values were recorded at the time of implant placement (baseline), at 8 weeks, and at 16 weeks using resonance frequency analysis (RFA). Cone-beam computed tomography (CBCT) scans were performed immediately after implant placement and at 16 weeks to measure marginal bone level changes at buccal, mesial, and distal aspects.

The primary outcome measure was implant stability, while the secondary outcome measure was marginal bone level change. The study aimed to test the hypothesis that local simvastatin application would enhance peri-implant bone healing, increase stability, and reduce marginal bone loss compared to the control group.

Ethical approval was obtained from the Research Ethics Committee, College of Dentistry, University of Baghdad, and all participants provided written informed consent before enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients ≥ 18 years of either gender.
2. Having missing teeth in maxillary jaw maxillary jaw( premolar and molar area) at least 6 months after teeth extraction.
3. Patients who had alveolar ridges of sufficient vertical and horizontal dimensions and were considered surgically straight forward cases according to SAC classification

Exclusion Criteria:

1. Patients with signs of acute or chronic infection in the implant zone
2. Patients with signs of parafunctional habits
3. Patients with history of systemic diseases or recent radiotherapy to the head and neck or chemotherapy.
4. Patients who had history or were currently under treatment with oral or intravenous bisphosphonate or statins other drugs that may alter bone metabolism
5. Patients who are heavy smoker or presented with severe periodontitis.
6. Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-07-06 (Actual); Study Completion 2025-07-06 (Actual)

PRIMARY OUTCOMES:
Implant Stability Quotient (ISQ) | Baseline, 8 weeks, and 16 weeks
  Implant stability was assessed using resonance frequency analysis (Osstell device). ISQ values were recorded at baseline (implant placement), 8 weeks, and 16 weeks postoperatively.

SECONDARY OUTCOMES:
Marginal Bone Level (MBL) | Baseline and 16 weeks
  Marginal bone level changes were measured radiographically using cone-beam computed tomography (CBCT) at baseline and 16 weeks, recorded at buccal, mesial, and distal aspects of the implant.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, University of Baghdad, Baghdad, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) or additional supporting documents will be shared. Data will remain confidential and stored securely at the College of Dentistry, University of Baghdad, in accordance with institutional ethical approval

REFERENCES:
- See also: Related Info — https://codental.uobaghdad.edu.iq/